CLINICAL TRIAL: NCT03601078
Title: A Phase 2, Multi-cohort, Open-label, Multicenter Study to Evaluate the Efficacy and Safety of bb2121 in Subjects With Relapsed and Refractory Multiple Myeloma and in Subjects With Clinical High-Risk Multiple Myeloma (KarMMa-2)
Brief Title: An Efficacy and Safety Study of bb2121 in Subjects With Relapsed and Refractory Multiple Myeloma and in Subjects With High-Risk Multiple Myeloma
Acronym: KarMMa-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB2121-MM-002; U1111-1216-4209 (Other: WHO); 2023-505183-10 (Other: EU CT Number)
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; bb2121; Relapsed and Refractory Multiple Myeloma; High Risk Multiple Myeloma; Phase 2; Multi-cohort; Open-label
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — idecabtagene vicleucel; Lenalidomide; talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: BB2121 in relapsed and refractory multiple myeloma participants (Experimental): bb2121 autologous CAR T cells will be infused at a dose ranging from 150 - 450 x 10^6 CAR+ T cells after receiving lymphodepleting chemotherapy
  Interventions: Biological: bb2121
- Cohort 1b: BB2121 with talquetamab in relapsed and refractory multiple myeloma participants (Experimental)
  Interventions: Biological: bb2121; Drug: Talquetamab
- Cohort 2a: BB2121 in multiple myeloma with Autologous stem cell transplantation participants (Experimental)
  Interventions: Biological: bb2121
- Cohort 2b: BB2121 in multiple myeloma without Autologous stem cell transplantation participants (Experimental)
  Interventions: Biological: bb2121
- Cohort 2c: BB2121 in multiple myeloma participants with inadequate response post ASCT (Experimental)
  Interventions: Biological: bb2121
- Cohort 3: BB2121 with lenalidomide maintenance in newly diagnosed multiple myeloma (Experimental)
  Interventions: Biological: bb2121; Drug: Lenalomide

INTERVENTIONS:
Biological: bb2121 — bb2121 consists of autologous T lymphocytes transduced with an anti-BCMA CAR lentiviral vector to express a chimeric antigen receptor targeting the human B cell maturation antigen (anti-BCMA CAR)
  Other Names: BMS-986395
Drug: Lenalomide — Specified dose on specified days
  Other Names: Revlimid®
  Arms: Cohort 3: BB2121 with lenalidomide maintenance in newly diagnosed multiple myeloma
Drug: Talquetamab — Specified dose on specified days
  Other Names: TALVEY
  Arms: Cohort 1b: BB2121 with talquetamab in relapsed and refractory multiple myeloma participants

SUMMARY:
This study is a multi-cohort, open-label, multicenter Phase 2 study to evaluate the efficacy and safety of bb2121 in participants with relapsed and refractory multiple myeloma (RRMM) (Cohort 1), in participants with RRMM who receive bridging therapy with talquetamab (Cohort 1b), in participants with multiple myeloma (MM) having progressed within 18 months of initial treatment with autologous stem cell transplantation (ASCT) (Cohort 2a) and without ASCT (Cohort 2b) or, in participants with inadequate response post ASCT during initial treatment (Cohort 2c) and the efficacy and safety of bb2121 used in combination with lenalidomide maintenance in participants with suboptimal response post ASCT (Cohort 3). Approximately 248 participants will be enrolled into one of three cohorts. Cohort 1 (including cohort 1b) will enroll approximately 126 RRMM subjects with ≥ 3 prior anti-myeloma treatment regimens. Cohort 2a will enroll approximately 39 MM subjects, with 1 prior anti-myeloma therapy including ASCT and with early relapse. Cohort 2b will enroll approximately 39 MM subjects with 1 prior anti-myeloma therapy not including ASCT and with early relapse. Cohort 2c will enroll approximately 30 MM subjects with inadequate response to ASCT during their initial anti-myeloma therapy. The cohorts will start in parallel and independently. Cohort 3 will enroll approximately 30 newly diagnosed multiple myeloma (NDMM) participants with suboptimal response to ASCT.

DETAILED DESCRIPTION:
Anti-myeloma bridging treatment is allowed for disease control while bb2121 is being manufactured for cohorts 1, 2a and 2b only. In Cohort 1b only, subjects will receive bridging therapy with 1 to 2 cycles of talquetamab, and initiate Lymphodepleting (LD) chemotherapy at least 14 days after the last dose of talquetamab.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF)
2. For Cohorts 1 and 2 only, participant has measurable disease, defined as:

   * M-protein (serum protein electrophoresis [sPEP] or urine protein electrophoresis [uPEP]): sPEP ≥ 0.5 g/dL or uPEP ≥ 200 mg/24 hours and/or
   * Light chain MM without measurable disease in the serum or urine: Serum immunoglobulin free light chain ≥ 10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio
3. Subjects with one of the following cohort specific requirements:

   Cohort 1 RRMM subjects with ≥ 3 prior anti-myeloma treatment regimens:
   * Subject must have received at least 3 prior anti-myeloma treatment regimens. Note: induction with or without hematopoietic stem cell transplant and with or without maintenance therapy is considered a single regimen
   * Subject must have undergone at least 2 consecutive cycles of treatment for each regimen, unless PD was the best response to the regimen
   * Subject must have received prior treatment with a proteasome inhibitor, an immunomodulatory agent and an anti-CD38 antibody
   * Subject has evidence of PD on or within 60 days of the most recent prior treatment regimen
   * Subject achieved a response (minimal response [MR] or better) to at least 1 prior treatment regimen

   Cohort 2 subjects with 1 prior anti-myeloma treatment regimen:
   * Subject must have received only 1 prior anti-myeloma treatment regimen. Note: induction with or without hematopoietic stem cell transplant and with or without maintenance therapy is considered a single regimen
   * Subject must have the following HR factors:
   * Early relapse defined as:

   Cohort 2a: PD < 18 months since date of start of initial therapy. Initial therapy must contain induction, ASCT (single or tandem) and lenalidomide containing maintenance.

   Cohort 2b: PD < 18 months since date of start or initial therapy which must contain at minimum, a proteasome inhibitor, an immunomodulatory agent and dexamethasone Cohort 2c: Subject must have received minimum 3 cycles of induction therapy which must contain at minimum, a proteasome inhibitor, an immunomodulatory agent and dexamethasone. Subjects must have had ASCT (single or tandem AND < VGPR (excluding PD) at first assessment between 70 to 110 days after last ASCT, with initial therapy without consolidation and maintenance.

   Cohort 3 participants with newly diagnosed MM (NDMM) who received only induction and ASCT, without subsequent consolidation or maintenance Cohort 3
   * Must have received 4 to 6 cycles of induction therapy which must contain at minimum, a proteasome inhibitor and an immunomodulatory agent and must have had single ASCT within 6 months prior to consent
   * Must have achieved documented PR or VGPR at first post-ASCT assessment approximately 100 days after ASCT and this response must be maintained at screening
   * Per Investigator's assessment, subject must be a candidate for single-agent lenalidomide maintenance
4. Subject must have Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
5. Subject must have recovery to Grade 1 or baseline of any non-hematologic toxicities due to prior treatments, excluding alopecia and Grade 2 neuropathy

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject used any investigational agents within 14 days prior to leukapheresis or, for Cohort 3, within 14 days prior to consent
2. Subject received any of the following within the last 14 days prior to leukapheresis or, for Cohort 3, within 14 days prior to consent:

   1. Plasmapheresis
   2. Major surgery (as defined by the investigator)
   3. Radiation therapy other than local therapy for myeloma associated bone lesions
   4. Use of any systemic anti-myeloma drug therapy
3. Subject with known central nervous system involvement with myeloma
4. Subject has clinical evidence of pulmonary leukostasis and disseminated intravascular coagulation
5. History or presence of clinically relevant central nervous system (CNS) pathology
6. Subject with active or history of plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome, or clinically significant amyloidosis
7. Inadequate organ function Subject with a history of Class III or IV congestive heart failure (CHF) or severe nonischemic cardiomyopathy, unstable or poorly controlled angina, myocardial infarction, or ventricular arrhythmia within the previous 6 months prior to starting study treatment
8. Ongoing treatment with chronic immunosuppressants
9. Previous history of an allogeneic hematopoietic stem cell transplantation or treatment with any gene therapy-based therapeutic for cancer or investigational cellular therapy for cancer or BCMA targeted therapy
10. Subject has received ASCT within 12 weeks prior to leukapheresis
11. Subject has history of primary immunodeficiency
12. Subject is positive for human immunodeficiency virus (HIV-1), chronic or active hepatitis B or active hepatitis A or C
13. Subject has uncontrolled systemic fungal, bacterial, viral or other infection (including tuberculosis) despite appropriate antibiotics or other treatment
14. Subject with prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 5 years
15. Pregnant or lactating women
16. Subject with known hypersensitivity to any component of bb2121 product, cyclophosphamide, fludarabine, and/or tocilizumab
17. Prior history of deep venous thrombosis (DVT) or pulmonary embolus (PE) within 6 months prior to consent (For Cohort 3)
18. For Cohort 1b, previous treatment with any G Protein-Coupled Receptor Class C Group 5 Member D (GPRC5D) targeted therapy or T-cell engagers
19. For Cohort 1b, known allergies, hypersensitivity, or intolerance to talquetamab or its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR)- Cohort 1 | Up to approximately 5 years (Participants will transition to the long term follow-up (LTFU) study after a minimum of 12 months post-infusion for Cohorts 1, 2a, 2b, and 2c; and after a minimum of 6 months post-infusion for Cohort 1b, at their next visit)
  Percentage of subjects who achieved partial response (PR) or better according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by the investigator
Complete response (CR) rate - Cohort 1b, 2a, 2b, 2c, and Cohort 3 | Up to approximately 5 years (Participants will transition to the LTFU study after a minimum of 12 months post-infusion for Cohorts 1, 2a, 2b, and 2c; and after a minimum of 6 months post-infusion for Cohort 1b, at their next visit)
  Percentage of subjects who achieved CR or stringent CR according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by the investigator

SECONDARY OUTCOMES:
Complete response (CR) rate - Cohort 1 | Up to approximately 5 years (Participants will transition to the LTFU study after a minimum of 12 months post-infusion for Cohorts 1, 2a, 2b, and 2c; and after a minimum of 6 months post-infusion for Cohort 1b, at their next visit)
  Percentage of subjects who achieved CR or better according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by the investigator
Overall response rate (ORR) - Cohort 1b, 2a, b, c and Cohort 3 | Up to approximately 5 years (Participants will transition to the LTFU study after a minimum of 12 months post-infusion for Cohorts 1, 2a, 2b, and 2c; and after a minimum of 6 months post-infusion for Cohort 1b, at their next visit)
  Percentage of subjects who achieved partial response (PR) or better according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by the investigator
Very good partial response (VGPR) rate - Cohort 2c | Up to approximately 5 years(Participants will transition to the LTFU study after a minimum of 12 months post-infusion for Cohorts 1, 2a, 2b, and 2c; and after a minimum of 6 months post-infusion for Cohort 1b, at their next visit)
  Percentage of subjects who achieved VGPR or better according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by the investigator
Time to response (TTR) | Up to approximately 5 years (Participants will transition to the LTFU study after a minimum of 12 months post-infusion for Cohorts 1, 2a, 2b, and 2c; and after a minimum of 6 months post-infusion for Cohort 1b, at their next visit)
  Time from first bb2121 infusion to first documentation of response (PR or greater) [Cohorts 1 and 2]; time from first dose of lenalidomide pre-leukapheresis to first documentation of response [Cohort 3 only]
Duration of response (DoR) | Up to approximately 5 years (Participants will transition to the LTFU study after a minimum of 12 months post-infusion for Cohorts 1, 2a, 2b, and 2c; and after a minimum of 6 months post-infusion for Cohort 1b, at their next visit)
  Time from first documentation of response (PR or greater) to first documentation of progressive disease (PD) or death from any cause, whichever occurs first
Progression-free survival (PFS) | Up to approximately 5 years (Participants will transition to the LTFU study after a minimum of 12 months post-infusion for Cohorts 1, 2a, 2b, and 2c; and after a minimum of 6 months post-infusion for Cohort 1b, at their next visit)
  Time from first bb2121 infusion to first documentation of PD, or death due to any cause, whichever occurs first (Cohorts 1 and 2); time from first dose of lenalidomide pre-leukapheresis to first documentation of PD, or death due to any cause, whichever occurs first (Cohort 3 only)
Time to progression (TTP) | Up to approximately 5 years (Participants will transition to the LTFU study after a minimum of 12 months post-infusion for Cohorts 1, 2a, 2b, and 2c; and after a minimum of 6 months post-infusion for Cohort 1b, at their next visit)
  Time from first bb2121 infusion to first documentation of PD (Cohorts 1 and 2); time from first dose of lenalidomide pre-leukapheresis to first documentation of PD (Cohort 3 only)
Overall survival (OS) | Up to approximately 5 years (Participants will transition to the LTFU study after a minimum of 12 months post-infusion for Cohorts 1, 2a, 2b, and 2c; and after a minimum of 6 months post-infusion for Cohort 1b, at their next visit)
  Time from first bb2121 infusion to time of death due to any cause (Cohorts 1 and 2); time from first dose of lenalidomide pre-leukapheresis to time of death due to any cause (Cohort 3 only)
Percentage of participants who received lenalidomide maintenance for the first 3 cycles following bb2121 infusion with at least 75% dose compliance - Cohort 3 | Up to 3 months
Pharmacokinetics - Cmax | Minimum 5 years after bb2121 infusion
  Maximum expansion of bb2121 chimeric antigen receptor (CAR) T cells
Pharmacokinetics - tmax | Minimum 5 years after bb2121 infusion
  Time to peak of bb2121 CAR T cells
Pharmacokinetics - AUC | Minimum 5 years after bb2121 infusion
  Area under the curve of CAR T cells
Pharmacokinetics - tlast | Minimum 5 years after bb2121 infusion
  Time to last measurable CAR T cells
Pharmacokinetics - AUC0-28days | Minimum 5 years after bb2121 infusion
  Area under the curve of CAR T cells from time zero to Day 28
Immunogenicity | Minimum of 2 years after bb2121 infusion
  Development of an anti-CAR antibody response
Subject-reported outcomes as measured by European Organization for Research and Treatment of Cancer Quality-of-Life questionnaire (EORTC-QLQ-C30) | Minimum 5 years after bb2121 infusion
  Questionnaire will be used as a measure of health-related quality of life
Subject-reported outcomes as measured by EuroQoL Group EQ-5D-5L Health Questionnaire | Minimum 5 years after bb2121 infusion
  Is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal
Subject-reported outcomes as measured by EORTC-QLQ-MY20 | Minimum 5 years after bb2121 infusion
  Is a 20-item myeloma module intended for use among patients varying in disease stage and treatment modality

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (25):
- United States (18):
  - Mayo Clinic in Arizona - Scottsdale, Scottsdale, Arizona
  - University Of California San Francisco Medical Center, San Francisco, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - University Of Nebraska, Omaha, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Mt Sinai Medical Center - NY, New York, New York
  - Columbia University Medical Center/New York-Presbyterian Hospital, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - University Of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center The University of Texas, Houston, Texas
  - Swedish Cancer Inst, Seattle, Washington
  - Froedtert Hospital BMT Medical College of Wisconsin, Milwaukee, Wisconsin
- Local Institution - 404, Poitiers, France
- Germany (2):
  - Local Institution - 506, Hamburg
  - Local Institution - 505, Würzburg
- Local Institution - 603, Bologna, Italy
- Spain (2):
  - Clinica Universidad de Navarra, Pamplona
  - Local Institution - 704, Salamanca
- Kings College Hospital NHS Foundation Trust, London, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT03601078.html